CLINICAL TRIAL: NCT05379634
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Nipocalimab in Participants With Active Idiopathic Inflammatory Myopathies
Brief Title: A Study of Nipocalimab in Participants With Active Idiopathic Inflammatory Myopathies
Acronym: SPIREA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR109210; 80202135IIM2001 (Other: Janssen Research & Development, LLC); 2023-505314-20-00 (Registry Identifier: EUCT number)
Expanded Access: NCT05221619 (Temporarily not available)
Record Dates: First submitted 2022-05-17; First posted 2022-05-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Myositis
MeSH Terms: conditions — Myositis | interventions — Glucocorticoids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nipocalimab (Experimental): Participants will receive Nipocalimab at Week 0 (Baseline) and then every 2 weeks (Q2W) up to Week 50 during double-blind period. Participants on glucocorticoids (GC) at baseline will receive a stable dose of oral GC (prednisone or equivalent) from 4 weeks prior to the first administration of study intervention to Week 0. No changes in GC doses are allowed between Week 0 and Week 24. From Week 24 to Week 44, GC doses will be tapered. No changes to GC doses will be allowed from Week 44 to Week 52. Eligible participants will enter long-term extension (LTE) period and continue receiving Nipocalimab starting from Week 52 up to Week 98 and will be followed up to Week 106.
  Interventions: Drug: Nipocalimab; Drug: Glucocorticoids
- Placebo (Placebo Comparator): Participants will receive Nipocalimab matching placebo at Week 0 (Baseline) and then Q2W up to Week 50 during double-blind period. Participants on GC at baseline will receive a stable dose of oral GC (prednisone or equivalent) from 4 weeks prior to the first administration of study intervention to Week 0. No changes in GC doses are allowed between Week 0 and Week 24. From Week 24 to Week 44, GC doses will be tapered. No changes to GC doses will be allowed from Week 44 to Week 52. Eligible participants will enter LTE period and will receive Nipocalimab treatment Q2W starting from Week 52 up to Week 98 and will be followed up to Week 106.
  Interventions: Other: Placebo; Drug: Glucocorticoids

INTERVENTIONS:
Drug: Nipocalimab — Nipocalimab will be administered intravenously in double-blind period and LTE period.
  Other Names: JNJ-80202135; JNJ-86507083
  Arms: Nipocalimab
Other: Placebo — Nipocalimab matching placebo will be administered intravenously in double-blind period.
  Arms: Placebo
Drug: Glucocorticoids — Prednisone or equivalent will be administered orally as Glucocorticoid.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Nipocalimab versus placebo in participants with active idiopathic inflammatory myopathies (IIM).

ELIGIBILITY:
Inclusion Criteria:

* Disease classification criteria: Participant meets the diagnostic criteria of probable or definite idiopathic inflammatory myopathies (IIM) based on 2017 The European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria for adult IIM at least 6 weeks prior to first administration of the study intervention
* If a participant is on regular or as needed treatment with low potency topical glucocorticoids (GC) that are allowed in the study or topical tacrolimus (TAC) to treat skin lesions, the dose and frequency should be stable for greater than or equal to (>=) 4 weeks prior to first administration of the study intervention as well as maintained at the same dose until Week 52 of the study
* Antibody positivity criteria: Any 1 of the myositis-specific antibodies (MSAs) positive: dermatomyositis (DM): anti-Mi-2 (Mi-2/nucleosome remodeling and deacetylase [NuRD] complex), anti-transcription intermediary factor 1-Gamma (TIF1-Gamma), anti- nuclear matrix protein 2 (NXP-2), anti-small ubiquitin-like modifier-1 activating enzyme; anti- antimelanoma differentiation-associated gene 5 (MDA-5) antibodies. Or immune-mediated necrotizing myopathy (IMNM): anti- signal recognition particle (SRP) and anti- 3-hydroxy-3-methylglutaryl-coenzyme A reductase (HMGCR) antibodies. Or anti-synthetase syndrome (ASyS): anti- histidyl- ribonucleic acid [tRNA] synthetase (Jo-1), anti- threonyl-tRNA synthetase (PL7), anti- alanyl-tRNA synthetase (PL12), anti- isoleucyl-tRNA synthetase (OJ), and anti- glycyl-tRNA synthetase (EJ) antibodies. If all MSAs are negative or more than 1 MSA is positive within different subtypes (defined by the central laboratory) at screening, the tests should be repeated during the screening period. If the same results are observed at retesting, the participant should not be enrolled in the study

Exclusion Criteria:

* Has a juvenile myositis diagnosis and now >=18 years old
* Has cancer-associated myositis defined as cancer diagnosis within 3 years of myositis diagnosis except for cervical carcinoma in situ and non-melanoma skin cancer (squamous cell carcinoma, basal cell carcinoma of the skin)
* Has comorbidities (example, asthma, chronic obstructive pulmonary disease [COPD]) which have required 3 or more courses of oral GC within 1 year prior to screening
* Has a history of primary immunodeficiency or secondary immunodeficiency not related to the treatment of the participants IIM
* Has experienced myocardial infarction (MI), unstable ischemic heart disease, or stroke within 12 weeks of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2026-09-16 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve at Least Minimal Improvement (Greater Than or Equal to [>=] 20) in IMACS TIS and on Less Than or Equal to (<=) 5 Milligrams per day (mg/day) of Oral Prednisone (or Equivalent) From Week 44 Through Week 52 | At Week 52
  Percentage of participants who achieve at least minimal improvement (>=20) in IMACS TIS at Week 52 and on <=5 mg/day of oral prednisone (or equivalent) from Week 44 through Week 52 will be reported. International Myositis Assessment and Clinical Studies Total Improvement Score (IMACS TIS) is a standardized clinical response criteria to assess minimal, moderate and major clinical improvement in adult participants with idiopathic inflammatory myopathies (IIM). Minimal improvement is defined as IMACS TIS greater than or equal to (>=) 20 in participants with IIM. The criteria use the 6 IMACS core set measures: physicians' global activity, patient global activity (PtGA), manual muscle testing (MMT)-8, muscle enzymes, myositis disease activity assessment tool (MDAAT), and health assessment questionnaire-disability index (HAQ-DI). The absolute percentage change in each measure with varying weights is combined to obtain a TIS on a scale of 0 to 100. Higher score indicates greater improvement.

SECONDARY OUTCOMES:
Percentage of Participants who Achieve at Least Minimal Improvement (>=20) in IMACS TIS | At Week 24
  IMACS TIS is a standardized clinical response criteria to assess minimal, moderate and major clinical improvement in adult participants with IIM. Minimal improvement is defined as IMACS TIS >=20 in participants with IIM. The criteria use the 6 IMACS core set measures: PhGA, PtGA, MMT-8, muscle enzymes, MDAAT, and HAQ-DI. The absolute percentage change in each measure with varying weights is combined to obtain a TIS on a scale of 0 to 100. Higher score indicates greater improvement.
IMACS TIS | At Week 52
  IMACS TIS is a standardized clinical response criteria to assess minimal, moderate and major clinical improvement in adult participants with IIM. The criteria use the 6 IMACS core set measures: PhGA, PtGA, MMT-8, muscle enzymes, MDAAT, and HAQ-DI. The absolute percentage change in each measure with varying weights is combined to obtain a TIS on a scale of 0 to 100. Higher score indicates greater improvement.
Percentage of Participants who Achieve at Least Moderate Improvement (>=40) in IMACS TIS | At Week 24
  IMACS TIS is a standardized clinical response criteria to assess minimal, moderate and major clinical improvement in adult participants with IIM. Moderate improvement is defined as IMACS TIS >=40 in participants with IIM. The criteria use the 6 IMACS core set measures: PhGA, PtGA, MMT-8, muscle enzymes, MDAAT, and HAQ-DI. The absolute percentage change in each measure with varying weights is combined to obtain a TIS on a scale of 0 to 100. Higher score indicates greater improvement.
Change From Baseline in Manual Muscle Testing (MMT)-8 at Week 52 | Baseline and Week 52
  Change from baseline in MMT-8 score at Week 52 will be reported. Manual muscle testing is a partially validated tool to assess muscle strength. It evaluates 8 muscle groups containing 1 axial, 5 proximal, and 2 distal muscle groups. MMT-8 score ranges from 0-150. Higher score indicates greater muscle strength, that is, less impairment of muscle.
IMACS TIS | At Week 24
  IMACS TIS is a standardized clinical response criteria to assess minimal, moderate and major clinical improvement in adult participants with IIM. The criteria use the 6 IMACS core set measures: PhGA, PtGA, MMT-8, muscle enzymes, MDAAT, and HAQ-DI. The absolute percentage change in each measure with varying weights is combined to obtain a TIS on a scale of 0 to 100. Higher score indicates greater improvement.
Percentage of Participants who Achieve at Least Moderate Improvement (>=40) in IMACS TIS | At Week 52
  IMACS TIS is a standardized clinical response criteria to assess minimal, moderate and major clinical improvement in adult participants with IIM. Moderate improvement is defined as IMACS TIS >=40 in participants with IIM. The criteria use the 6 IMACS core set measures: PhGA, PtGA, MMT-8, muscle enzymes, MDAAT, and HAQ-DI. The absolute percentage change in each measure with varying weights is combined to obtain a TIS on a scale of 0 to 100. Higher score indicates greater improvement.
Percentage of Participants who Achieve at Least Major Improvement (>=60) in IMACS TIS | At Weeks 24 and 52
  IMACS TIS is a standardized clinical response criteria to assess minimal, moderate and major clinical improvement in adult participants with IIM. Major improvement is defined as IMACS TIS >=60 in participants with IIM. The criteria use the 6 IMACS core set measures: PhGA, PtGA, MMT-8, muscle enzymes, MDAAT and HAQ-DI. The absolute percentage change in each measure with varying weights is combined to obtain a TIS on a scale of 0 to 100. Higher score indicates greater improvement.
Change From Baseline in MMT-8 at Week 24 | Baseline and Week 24
  Change from baseline in MMT-8 score at Week 24 will be reported. Manual Muscle Testing is a partially validated tool to assess muscle strength. It evaluates 8 muscle groups containing 1 axial, 5 proximal, and 2 distal muscle groups. MMT-8 score ranges from 0-150. Higher score indicates greater muscle strength, that is, less impairment of muscle.
Change From Baseline in Physician Global Assessment (PhGA) at Weeks 24 and Week 52 | Baseline, Weeks 24 and 52
  Change from baseline in PhGA at Weeks 24 and 52 will be reported. Physician Global Activity is a partially validated tool to measure the global evaluation by the physician of the participant's overall disease activity at the time of assessment using a 10 centimeter (cm) visual analogue scale (VAS), where 0 cm= no evidence of disease activity and 10 cm= extremely active or severe disease activity.
Change From Baseline in Extramuscular Global Assessment (Myositis Disease Activity Assessment Tool [MDAAT]) at Weeks 24 and 52 | Baseline, Weeks 24 and 52
  Change from baseline in MDAAT score at Weeks 24 and 52 will be reported. This is a validated tool which measures the degree of disease activity of extramuscular organ systems and muscle. MDAAT is scored on a 10 centimeter (cm) scale ranging from 0-10 cm where, 0 cm = absent and 10 cm = maximum disease activity. Higher score indicates more disease activity.
Change From Baseline in Serum Muscle Enzymes Levels at Weeks 24 and 52 | Baseline, Weeks 24 and 52
  Change from baseline in serum muscle enzymes levels (creatine kinase [CK], alanine aminotransferase [ALT], aspartate aminotransferase [AST], lactate dehydrogenase [LDH], and aldolase) at Weeks 24 and 52 will be reported.
Percentage of Participants who Achieve Oral Glucocorticoids (GC) Reduction to 5 Milligrams per day (mg/day) of Oral Prednisone (or Equivalent), Among Participants on Oral GC Greater Than (>) 5 mg/day at Baseline | From Week 44 through Week 52
  Percentage of participants who achieve oral GC reduction to 5 mg/day of oral prednisone (or equivalent) at Week 44 and maintain that reduction through Week 52, among participants on oral GC >5 mg/day at baseline will be reported.
Percentage of Participants who Achieve at Least Minimal Improvement (>=20) in IMACS TIS From Week 44 Through Week 52 and on Less Than or Equal to (<=) 5 mg/day of Oral Prednisone (or Equivalent) From Week 44 Through Week 52 | From Week 44 through Week 52
  Percentage of participants who achieve at least minimal improvement (>=20) in IMACS TIS from Week 44 through Week 52 and on <=5 mg/day of oral prednisone (or equivalent) from Week 44 through Week 52 will be reported. IMACS TIS is a standardized clinical response criteria to assess minimal, moderate and major clinical improvement in adult participants with IIM. Minimal improvement is defined as IMACS TIS >=20 in participants with IIM. The criteria use the 6 IMACS core set measures: PhGA, PtGA, MMT-8, muscle enzymes, MDAAT, and HAQ-DI. The absolute percentage change in each measure with varying weights is combined to obtain a TIS on a scale of 0 to 100. Higher score indicates greater improvement.
Percentage of Participants on <=5 mg/day of Oral Prednisone (or Equivalent) From Week 44 Through Week 52 | From Week 44 through Week 52
  Percentage of participants on <=5 mg/day of oral prednisone (or equivalent) from Week 44 through Week 52 will be reported.
Percentage of Participants who Achieve At Least Minimal Improvement (>=20) in IMACS TIS and Achieve Oral GC Reduction to 5 mg/day at Week 44 and Maintain That Reduction Through Week 52, Among Participants on Oral GC >5 mg/day at Baseline | From Week 44 through Week 52
  Percentage of participants who achieve at least minimal improvement (>=20) in IMACS TIS from Week 44 through Week 52 and achieve oral GC reduction to 5 mg/day of prednisone (or equivalent) at Week 44 and maintain that reduction through Week 52, among participants on oral GC >5 mg/day at baseline will be reported. IMACS TIS is a standardized clinical response criteria to assess minimal, moderate and major clinical improvement in adult participants with IIM. Minimal improvement is defined as IMACS TIS >=20 in participants with IIM. The criteria use the 6 IMACS core set measures: PhGA, PtGA, MMT-8, muscle enzymes, MDAAT, and HAQ-DI. The absolute percentage change in each measure with varying weights is combined to obtain a TIS on a scale of 0 to 100. Higher score indicates greater improvement.
Percentage of Participants who Achieve at Least Minimal Improvement (>=20) in IMACS TIS From Week 44 Through Week 52 and on <=7.5 mg/day of Oral Prednisone (or Equivalent) From Week 44 Through Week 52 | From Week 44 through Week 52
  Percentage of participants who achieve at least minimal improvement (>=20) in IMACS TIS from Week 44 through Week 52 and on <=7.5 mg/day of Oral Prednisone (or Equivalent) from Week 44 through Week 52 will be reported. IMACS TIS is a standardized clinical response criteria to assess minimal, moderate and major clinical improvement in adult participants with IIM. Minimal improvement is defined as IMACS TIS >=20 in participants with IIM. The criteria use the 6 IMACS core set measures: PhGA, PtGA, MMT-8, muscle enzymes, MDAAT, and HAQ-DI. The absolute percentage change in each measure with varying weights is combined to obtain a TIS on a scale of 0 to 100. Higher score indicates greater improvement.
Percentage of Participants who Achieve Oral GC Reduction to <=7.5 mg/day of Oral Prednisone (or Equivalent) at Week 44 and Maintain That Reduction Through Week 52, Among Participants on Oral GC >7.5 mg/day at Baseline | At Week 44 through Week 52
  Percentage of participants who achieve oral GC reduction to <=7.5 mg/day of oral prednisone (or equivalent) at Week 44 and maintain that reduction through Week 52, among participants on oral GC >7.5 mg/day at baseline will be reported.
Percentage of Participants who Achieve at Least Minimal Improvement (>=20) in IMACS TIS and Achieve Oral GC Reduction to <=7.5 mg/day at Week 44 and Maintain That Reduction Through Week 52, Among Participants on Oral GC >7.5 mg/day at Baseline | From Week 44 through Week 52
  Percentage of participants who achieve at least minimal improvement (>=20) in IMACS TIS from Week 44 through Week 52 and achieve oral GC reduction to <=7.5 mg/day of oral prednisone (or equivalent) at Week 44 and maintain that reduction through Week 52, among participants on oral GC >7.5 mg/day at Baseline will be reported. IMACS TIS is a standardized clinical response criteria to assess minimal, moderate and major clinical improvement in adult participants with IIM. Minimal improvement is defined as IMACS TIS >=20 in participants with IIM. The criteria use the 6 IMACS core set measures: PhGA, PtGA, MMT-8, muscle enzymes, MDAAT, and HAQ-DI. The absolute percentage change in each measure with varying weights is combined to obtain a TIS on a scale of 0 to 100. Higher score indicates greater improvement.
IMACS TIS Over Time | Up to 106 weeks
  IMACS TIS is a standardized clinical response criteria to assess minimal, moderate and major clinical improvement in adult participants with IIM. The criteria use the 6 IMACS core set measures: PhGA, PtGA, MMT-8, muscle enzymes, MDAAT, and HAQ-DI. The absolute percentage change in each measure with varying weights is combined to obtain a TIS on a scale of 0 to 100. Higher score indicates greater improvement.
Change From Baseline in the Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) Scale Score at Weeks 24 and 52 | Baseline, Weeks 24 and 52
  The CDASI scale is a validated dermatomyositis (DM) specific instrument that systematically quantifies activity and damage in the skin of participant with DM. Disease involvement in 15 different anatomical locations is rated using three activity scales (erythema, scale, erosion/ulceration) and two damage measures (poikiloderma, calcinosis) measures. Gottron's papules/sign on the hands are also evaluated in terms of activity (erythema/ulceration) and damage (dyspigmentation or scarring). Disease activity scores range from 0 to 100. Higher scores indicate greater disease activity.
Change in CDASI Scale Score Over Time | Up to 106 Weeks
  The CDASI scale is a validated DM specific instrument that systematically quantifies activity and damage in the skin of participant with DM. Disease involvement in 15 different anatomical locations is rated using three activity scales (erythema, scale, erosion/ulceration) and two damage measures (poikiloderma, calcinosis) measures. Gottron's papules/sign on the hands are also evaluated in terms of activity (erythema/ulceration) and damage (dyspigmentation or scarring). Disease activity scores range from 0 to 100. Higher scores indicate greater disease activity.
Percentage of Participants With Treatment-Emergent Adverse Events (AEs) | Up to 106 weeks
  Any AE occurring at or after the initial administration of study intervention through the safety follow-up visit will be considered as treatment-emergent. An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product that does not necessarily have a causal relationship with the intervention.
Percentage of Participants With Treatment-Emergent Serious Adverse Events (SAEs) | Up to 106 weeks
  Any AE occurring at or after the initial administration of study intervention through the safety follow-up visit will be considered as treatment-emergent. An SAE is any untoward medical occurrence that at any dose: results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS)- Physical Function (PF)-20 | Baseline and Week 52
  PROMIS-PF-20 is a participant self-administered 20-item questionnaire assessing the physical function domain. It includes 14 items regarding patients' ability to conduct specific functional activities and 6 items regarding the extent to which their health limits their ability to perform a range of physical activities currently. The 5-point response options for the former items range from 1 "Unable to do" to 5 "Without any difficulty" and the latter items range from 1 "Cannot do" to 5 "Not at all" with higher scores indicating better functioning. The overall score ranges from 0 to 100, where higher score indicates better physical function.
Change From Baseline in Functional Disability Using the Health Assessment Questionnaire-disability Index (HAQ-DI) | Baseline, Weeks 24 and 52
  HAQ-DI score assess functional status of participant. It is 20 question instrument that assess degree of functional disability a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and common activities of daily living). Responses in each functional area are scored from 0=indicating no difficulty, to 3=indicating inability to perform a task in that area. Total HAQ score is average of the computed categories scores ranging from 0-3 where 0=least difficulty and 3=extreme difficulty. Lower scores are indicative of better functioning.
Serum Nipocalimab Concentration Over Time | Baseline Up to Week 98
  Serum nipocalimab concentration over time will be reported. Serum nipocalimab concentration will be derived using population pharmacokinetic (PK) modeling.
Number of Participants With Anti-drug Antibody (ADA) Measured Using a Validated, Specific, and Sensitive Immunoassay Method | Baseline Up to Week 106
  Number of participants with ADA to Nipocalimab measured using a validated, specific, and sensitive immunoassay method will be reported.
Number of Participants With Neutralizing Antibodies (Nabs) to Nipocalimab Measured Using a Validated, Specific, and Sensitive Immunoassay Method | Baseline Up to Week 106
  Number of participants with Nabs to Nipocalimab measured using a validated, specific, and sensitive immunoassay method will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (57):
- United States (19):
  - Arizona Arthritis and Rheumatology Research PLLC, Phoenix, Arizona
  - HonorHealth Neurology, Scottsdale, Arizona
  - Attune Health Autoimmune and Inflamation Care and Research, Beverly Hills, California
  - University of California Irvine Medical Center, Orange, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - FM Clinical Research, LLC South Florida Neurology Associates, P. A., Boca Raton, Florida
  - Integral Rheumatology And Immunology Specialists, Plantation, Florida
  - University of South Florida, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - The Brigham and Women's Hospital, Inc., Boston, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Saint Clair Shores, Michigan
  - Wexner Medical Center at the Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania - Perelman School of Medicine, Philadelphia, Pennsylvania
  - ACME Research Arthritis and Osteoporosis Center, Orangeburg, South Carolina
  - Nervie and Muscle Center of Texas, Houston, Texas
  - University of Texas at Houston Medical School, Houston, Texas
- Canada (2):
  - Lawson Health Research / London Health Sciences Center Research, London, Ontario
  - AMIR Research, Montreal, Quebec
- Revmatologicky ustav, Prague, Czechia
- France (3):
  - Hospital Pasteur, Nice
  - Hôpital Pitié-Salpétrière, Paris
  - Nouvel Hopital Civil, Strasbourg
- Germany (3):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Klinikum der Universitaet Muenchen, München
  - Immanuel Klinik Rüdersdorf, Rüdersdorf Bei Berlin
- Hungary (2):
  - Orszagos Mozgasszervi Intezet ORFI Campus, Budapest
  - Debreceni Egyetem, Debrecen
- Italy (4):
  - A.O. Universitaria Ospedali Riuniti di Ancona, Ancona
  - IRCSS Ospedale San Raffaele Turro, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
- Japan (9):
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - St Marianna University Hospital, Kanagawa
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano
  - Tokushukai Chiba-Nishi General Hospital, Matsudo-shi
  - Shinshu University Hospital, Matsumoto
  - Tohoku University Hospital, Sendai
  - St. Luke's International Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
- Mexico (4):
  - Centro Integral en Reumatologia S A de C V, Guadalajara
  - Centro de Estudios de Investigacion Basica y Clinica, S.C., Guadalajara
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - CITER Centro de Investigacion y Tratamiento de las Enfermedades Reumaticas S A de C V, México
- Poland (2):
  - Szpital Uniwersytecki nr 2 im dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Narodowy Instytut Geriatrii Reumatologii i Rehabilitacji im prof dr hab med Eleonory Reicher, Warsaw
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (3):
  - Hosp. Univ. de Bellvitge, Barcelona
  - Hosp. Univ. de La Paz, Madrid
  - Hosp. Univ. Marques de Valdecilla, Santander
- United Kingdom (3):
  - Western General Hospital, Edinburgh
  - University College London Hospitals NHSFT, London
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency